CLINICAL TRIAL: NCT00490178
Title: An Open Label, Multicenter Trial Assessing the Acceptability of a New Fixed Combination of Fenofibrate 80 mg BID and Metformin 1000 mg BID in Patients With Type 2 Diabetes and Dyslipidemia
Brief Title: Acceptability Study of a New Fixed Combination of Fenofibrate 80 mg BID and Metformin 1000 mg BID in Type 2 Diabetes and Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C LF23-0121 06 02; 2006-002848-28
Record Dates: First submitted 2007-06-21; First posted 2007-06-22 (Estimated); Last update posted 2007-09-03 (Estimated); Status verified 2007-08

CONDITIONS: Diabetes Mellitus, Type 2; Dyslipidemia
Keywords: Type II diabetes; dyslipidemia; metformin; fenofibrate; synordia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias | interventions — Fenofibrate; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fenofibrate 80 mg and metformin 1000 mg (fixed combination)

SUMMARY:
The present study aims to assess the acceptability of a 4 week treatment of a new fixed-dose combination of fenofibrate and metformin, in patients with type 2 diabetes and dyslipidemia

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged from 20 to 80 years (at inclusion visit).
2. Type 2 diabetes treated with a stable dose of metformin for a minimum of 3 months either alone or in combination with another oral hypoglycaemic agent.
3. Dyslipidemia treated with 160 mg fenofibrate (or bioequivalent formulations) for a minimum of 3 months either alone or in combination with a statin.
4. And having signed a written informed consent.-

Exclusion Criteria:

1. Known Type 1 Diabetes, uncontrolled type 2 diabetes [HbA1c > 9.5 %, Fasting plasma glucose (FPG) > 240 mg/dL (> 13.4 mmol/L) on the last performed blood sample (within the last 3 months)].
2. TG > 500 mg/dL (> 5.65 mmol/L) on the last performed blood sample (within the last 3 months).
3. Women who are not surgically sterilized (i.e. bilateral tubal ligation, bilateral or two unilateral oophorectomies, hysterectomy) or not using adequate contraceptive methods (i.e. oral contraceptives, approved hormonal implant, intrauterine device, diaphragm with spermicide, condom with spermicide) or not postmenopausal (> 1 year since their last menstrual period).
4. Pregnant or lactating women.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (3):
- France (3):
  - Site 3, Marseille
  - Site 1, Nantes
  - Site 2, Tours